CLINICAL TRIAL: NCT05211739
Title: Clinical Assessment of a Daily Wear Monthly Replacement Silicone Hydrogel Toric Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLV201-C002
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Refractive Errors; Astigmatism
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID205255 Toric, then Biofinity Toric (Other): Lehfilcon A toric contact lenses worn first, with comfilcon A toric contact lenses worn second, as randomized. Each product will be worn bilaterally (in both eyes) during waking hours for at least 5 days per week, with up to 10-12 hours wear time per day over a 30-day period. CLEAR CARE will be used for nightly contact lens cleaning and disinfection.
  Interventions: Device: Lehfilcon A toric contact lenses; Device: Comfilcon A toric contact lenses; Device: CLEAR CARE
- Biofinity Toric, then LID205255 Toric (Other): Comfilcon A toric contact lenses worn first, with lehfilcon A toric contact lenses worn second, as randomized. Each product will be worn bilaterally (in both eyes) during waking hours for at least 5 days per week, with up to 10-12 hours wear time per day over a 30-day period. CLEAR CARE will be used for nightly contact lens cleaning and disinfection.
  Interventions: Device: Lehfilcon A toric contact lenses; Device: Comfilcon A toric contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A toric contact lenses — FDA-cleared silicone hydrogel toric contact lenses used as indicated
  Other Names: LID205255 Toric
Device: Comfilcon A toric contact lenses — Commercially available silicone hydrogel toric contact lenses used as indicated
  Other Names: Biofinity Toric; CooperVision® Biofinity® Toric
Device: CLEAR CARE — Hydrogen peroxide-based contact lens cleaning and disinfecting solution

SUMMARY:
The purpose of this clinical study is to assess the clinical performance of an investigational toric soft contact lens compared to a commercially available toric contact lens in a crossover dispense trial when worn in a daily wear modality for 30 days, each study lens type.

DETAILED DESCRIPTION:
Subjects will be randomized to 1 of 2 crossover wear sequences. Subjects will be expected to attend 5 office visits, for a total individual duration of participation in the study of approximately 60 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wearers of weekly/monthly toric soft contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months;
* Best corrected distance visual acuity (as determined by manifest refraction at screening) better than or equal to 20/25 Snellen in each eye.
* Able to wear contact lenses within the range of available sphere & cylinder power and axes.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Daily disposable contact lens wearers.
* Monovision and multifocal contact lens wearers.
* Habitual Biofinity Toric/Biofinity Toric XR contact lens wearers in the past 3 months prior to consent.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (7):
- United States (7):
  - Sabal Eye Care, Longwood, Florida
  - Drs. Giedd, P.A., Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Kannarr Eye Care LLC, Pittsburg, Kansas
  - Fischer Laser Eye Center, Willmar, Minnesota
  - SUNY College of Optometry Clinical Vision Research Center, New York, New York
  - West Bay Eye Associates, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 7 investigative sites located in the United States.
Pre-assignment Details: Of the 76 subjects enrolled in the study (i.e., signed informed consent), 2 subjects were exited prior to randomization as screen failures, and 1 randomized subject withdrew prior to exposure to the study lenses. This reporting group includes all randomized subjects/eyes (74/148).
Units Other Than Participants: eyes
Groups:
- LID205255 Toric, Then Biofinity Toric: Lehfilcon A toric contact lenses worn first, with comfilcon A toric contact lenses worn second, as randomized. Each product was worn bilaterally (in both eyes) during waking hours for at least 5 days per week, with up to 10-12 hours wear time per day over a 30-day period. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
- Biofinity Toric, Then LID205255 Toric: Comfilcon A toric contact lenses worn first, with lehfilcon A toric contact lenses worn second, as randomized. Each product was worn bilaterally (in both eyes) during waking hours for at least 5 days per week, with up to 10-12 hours wear time per day over a 30-day period. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
Period: First Wear Period (Approx 30 Days)
Arm/Group | LID205255 Toric, Then Biofinity Toric | Biofinity Toric, Then LID205255 Toric
Started | 36; 72 eyes | 38; 76 eyes
Exposed to Study Lenses | 35; 70 eyes | 38; 76 eyes
Completed | 35; 70 eyes | 36; 72 eyes
Not Completed | 1; 2 eyes | 2; 4 eyes
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject Prior to Exposure to the Study Lenses | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Wear Period (Approx 30 Days)
Arm/Group | LID205255 Toric, Then Biofinity Toric | Biofinity Toric, Then LID205255 Toric
Started | 35; 70 eyes | 36; 72 eyes
Completed | 34; 68 eyes | 36; 72 eyes
Not Completed | 1; 2 eyes | 0; 0 eyes
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID205255 Toric, Then Biofinity Toric | Biofinity Toric, Then LID205255 Toric | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: year] | 32.9 (8.3) | 35.8 (10.2) | 34.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 32 | 63
  Black or African American | 2 | 3 | 5
  Asian | 3 | 2 | 5
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) With Study Lenses
Description: Visual acuity (VA) was collected for each eye individually with study lenses in place using a letter chart. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity. No inferences were pre-specified for the primary effectiveness endpoint; therefore, no hypothesis testing was performed.
Time Frame: Day 1 and Day 30, each wear period (approximately 30 days)
Population: All subjects exposed to any study lenses evaluated in this study, as randomized, with non-missing data at the respective visit.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID205255 Toric: Lehfilcon A toric contact lenses worn first or second, as randomized, in both eyes during waking hours for at least 5 days per week, with up to 10-12 hours wear time per day over a 30-day period. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
- Biofinity Toric: Comfilcon A toric contact lenses worn first or second, as randomized, in both eyes during waking hours for at least 5 days per week, with up to 10-12 hours wear time per day over a 30-day period. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
Arm/Group | LID205255 Toric | Biofinity Toric
Number analyzed (Participants) | 71 | 73
Number analyzed (eyes) | 142 | 146
logMAR
  Day 1 | -0.06 (0.09) | -0.07 (0.09)
  Day 30: number analyzed (Participants) | 71 | 70
  Day 30: number analyzed (eyes) | 142 | 140
  Day 30 | -0.08 (0.09) | -0.06 (0.08)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 60 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID205255 Toric Ocular; LID205255 Toric Nonocular: Events reported in this group occurred while exposed to the lehfilcon A toric contact lenses
- Biofinity Toric Ocular; Biofinity Toric Nonocular: Events reported in this group occurred while exposed to the comfilcon A toric contact lenses
Arm/Group | Pretreatment | LID205255 Toric Ocular | LID205255 Toric Nonocular | Biofinity Toric Ocular | Biofinity Toric Nonocular
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/142 | 0/71 | 0/146 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/142 | 0/71 | 0/146 | 0/73
Other Adverse Events (participants affected / at risk) | 0/73 | 0/142 | 0/71 | 0/146 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT05211739/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05211739/SAP_001.pdf